CLINICAL TRIAL: NCT02934438
Title: The Effects of an Oral Nitric Oxide Lozenge on Peripheral Artery Disease
Brief Title: Effect of Neo40 on PAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HumanN (Industry)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R41AT009171-01A1 (NIH)
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Peripheral Artery Disease
Keywords: nitric oxide; Neo40 supplement,; exercise tolerance
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neo40 Supplement (Active Comparator): Utilizing intellectual property developed out of the University of Texas Health Science Center in Houston, Neo40 is a GMP certified, over the counter, all natural formulation that provides a system for generating NO in an endothelium-dependent and independent manner. The NEO40™ Daily™ product ingredients list and packaging was submitted to FDA Office of Compliance by Neogenis Labs, Inc. for use as a dietary supplement. It is made up of Beet root extract, hawthorne berry, Vitamin C, L-citrulline and sodium nitrite. The lozenges utilize natural product chemistry activated by the saliva to generate authentic NO gas in the oral cavity through the one-electron reduction of nitrite. This product's formulation was designed to be a quick dissolve that melts in the mouth within four to five minutes.
  Interventions: Dietary Supplement: Neo40
- Placebo (Placebo Comparator): A placebo product has been manufactured that looks, tastes and feels like the Neo40 active lozenge without the active ingredients
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Neo40
  Arms: Neo40 Supplement
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Reduced nitric oxide (NO) availability is a hallmark of a number of cardiovascular diseases (CVD) including peripheral artery disease (PAD). The investigators will test the hypothesis that sub-chronic NEO40™ supplementation will improve vascular NO function and improve intermittent claudication in patients with PAD. Using a prospective, double blind, placebo controlled experimental design in 30 patients, graded treadmill tests will be performed at baseline and after 3 months after randomization, according to the Skinner-Gardner protocol. Initial claudication distance (ICD) and absolute claudication distance (ACD) will be recorded. Two consecutive treadmill tests will be performed within 1 week at baseline (before administration of study drug); and 2 test will be performed at 3 months. Functional status will also be assessed by the Walking Impairment Questionnaire and the Health Status Survey SF-36 questionnaire (SF-36). Vascular function will be assessed with the use of a Vendys® vascular reactivity (endothelial function) test (Endothelix Inc). Digital pulse amplitude will be assessed using sensor probes on the index finger during reactive hyperemia. Blood will be collected for measurement (by Neogenis) of plasma levels of nitrite and nitrate at baseline and at the completion of the study. Based on previously published trials using this NO technology, the investigators predict that the group receiving the active supplement will exhibit an improvement in claudication distance and all measures of vascular function after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Persons of at least 45 years of age
* Persons with unilateral or bilateral PAD confirmed by a resting ankle-brachial index (ABI) <0.9
* Persons with stable intermittent claudication for the previous 3 months
* Persons with the ability to walk 1 to 12 minutes on a treadmill. The pre-randomization treadmill test is limited by exercise-induced leg pain, which is relieved by cessation of the test. Variability of maximum walking distances between 2 consecutive screening treadmill tests will be <10%.

Exclusion Criteria:

* Persons with ischemic rest pain, ulceration or gangrene
* Persons with history in the previous 3 months of acute coronary syndrome or revascularization involving the peripheral or coronary arteries
* Persons with major amputation
* Persons with malignancy within the previous 5 years (except for treated non-melanoma skin cancer)
* Persons with proliferative retinopathy
* Persons with uncontrolled hypertension
* Persons with active inflammatory, infectious, or autoimmune diseases.
* Persons taking taking phosphodiesterase inhibitors, organic nitrates and/or hydralazine

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Skinner-Gardner treadmill protocol. | 3 months
  The primary end point is the change at 3 months in the absolute claudication distance. Distance will be measured in meters walked on treadmill

SECONDARY OUTCOMES:
Endothelial function | 3 months
  Secondary objectives are to evaluate endothelial function. EndoPAT score of 1.67 and below correlates to endothelial dysfunction.

IPD SHARING:
Plan to Share IPD: Undecided